CLINICAL TRIAL: NCT05254093
Title: The Analgesic Effect of Single Shot Anterior Quadratus Lumborum Block Versus Erector Spinae Plane Block After Elective Cesarean Section: A Randomized Controlled Douple Blinded Trial
Brief Title: Anterior Quadratus Lumborum Block Versus Erector Spinae Plane Block After Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, Principal Investigator, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-60-2021
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Cesarean Section; Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (No Intervention)
- group B (Active Comparator)
  Interventions: Other: Quadratus lumborum block
- group C (Active Comparator)
  Interventions: Other: erector spinae plane block

INTERVENTIONS:
Other: Quadratus lumborum block — quadratus lumborum block, anterior approach using a curvilinear (5-8MHz) transducer. The transducer will be positioned transverse above the iliac crest at the posterior axillary line and slided posteriorly till the Shamrock sign is identified (the transvers process represent the stem and the attached erector spinae, QL and Psoas major muscles represent the three leaves). A 22 G, 100 mm needle will be advanced in-plane from lateral to medial through the QL muscle to reach the inter-fascial plane between the QL and psoas major muscles, posterior to the transversalis fascia. After ensuring negative aspiration, the local anesthetic solution (20 ml of 0.25% isobaric bupivacaine) will be injected anterior to the QL muscle. The procedure will be repeated on the opposite side of the back
  Arms: group B
Other: erector spinae plane block — the block will be given at the level of the 9th thoracic transverse process using a linear 6-13 MHz ultrasound transducer. The transducer will be positioned vertically 3 cm to the side of the midline to visualize the muscles of the back, the transverse process, and the pleura between the two transverse processes. Then, a 22G 10-mm needle will be introduced in the cranial-caudal direction toward the transverse process (T9) using the in-plane method till the needle tip crosses all the muscles. The tip of needle should be in the plane between the transverse process and the erector spinae muscle. After ensuring negative aspiration, the local anesthetic solution (20 ml of 0.25% isobaric bupivacaine) will be injected below the muscle. The procedure will be repeated on the opposite side of the back
  Arms: group C

SUMMARY:
Cesarean section is the one of the most common surgical procedures. Inadequate pain management is associated with increased morbidity, costs, and maternal dissatisfaction. Furthermore, effective postoperative pain management enables mothers to care for their newborn infants. Systemic and neuraxial opioids are the cornerstone of postoperative pain management; however, opioids are associated with significant side effect such as respiratory depression, urine retention, constipation, and itching. To reduce the postoperative opioids requirement and subsequently their side effects, multimodal regimen is advice including neuraxial anesthesia, neuraxial morphine, regular administration of non-opioids analgesia (non-steroidal anti-inflammatory drugs and acetaminophen) and planned use of opioid for breakthrough pain.

The addition of peripheral nerve blocks to the multimodal analgesic plan was found to reduced postoperative opioids requirement in non-obstetric procedures.

Quadratus lumborum (QLB) and erector spinae plane (ESPB) blocks are relatively new techniques for peripheral nerve block and showed promising results in managing pain after Cesarean delivery.

There are several types of QLB that had been described. Lateral (QLB1), posterior (QLB2), and anterior (QLB3) quadratus lumborum blocks been studied in cesarean delivery and were found to reduce opioids requirement when compared against placebo. Cadaver studies suggest that local anesthetic deposition at QLB1 diffuses mainly to the transversus abdominis muscle plane while, at QLB2, and at QLB3 spread may occur into the thoracic paravertebral space providing additional visceral pain control.

ESPB can provide both visceral and somatic analgesia due to anterior spread to the paravertebral space. ESPB was found to reduce postoperative opioids requirement in comparison to transversus abdominis plane block and intrathecal morphine.

To the best of our knowledge, there is no published data comparing the analgesic effect of QLB3 (anterior QL) and ESPB after elective cesarean delivery.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and pre-medication drugs will be delivered (metoclopramide 10 mg, and ranitidine 50 mg). Lactated Ringer's co-load will be rapidly infused at a rate of 15 mL.Kg-1 over 10 minutes.

Spinal anesthesia will be achieved by injecting 2.0 to 2.3 mg hyperbaric bupivacaine 0.5% plus 25 mcg fentanyl in L3-L4 or L4-L5 interspace.

The spinal block will be performed in the sitting position using a 25G spinal needle through midline approach. The participant will be then positioned supine with left-lateral uterine tilt. Pinprick was used for evaluation of block success 5 minutes after intrathecal injection. Successful block was confirmed if sensory block level was at T4 at least.

After skin closure and the covering of the wound with a dressing, patients received intravenous paracetamol (1 g) and ketorolac (30 mg).

Spinal block height will be assessed at the end of surgery to ensure enough anesthesia at the site of block performance. If the site of needle entry was not anesthetized, a local infiltration with 2ml of 20% lidocaine will be injected prior to the block. Patients will be blinded to block allocation using the surgical drapes to occlude their view. The patient will be into the lateral position and the back will be prepared in an aseptic manner.

after the end of the procedure the patients will receive their assigned intervention The blocks will be performed by experienced operator who will be informed of the patient group after patient positioning. The patient and the assessor of the block will be blinded to the study group.

Postoperative care All patients will receive parenteral paracetamol 1 g/6hours and ketorolac 30 mg/8hours postoperatively. Pain assessments using numerical rate scale (NRS) will be performed at rest and during movement (knee flexion) at 0.5, 1, 2, 4, 6, 18, 24 h after leaving the operating room. If NRS score is > 3 intravenous titration of 2 mg morphine given slowly to be repeated after 30 minutes if pain persisted. if other opioid given, the morphine equivalent dose will be calculated from the opioid conversion chart.

All scores will be assigned by each patient with the assistance of an anesthesiologist not responsible for the surgical intervention.

Intravenous ondansetron 4 mg will be given to treat nausea or vomiting. Complications: nausea, vomiting, itching, urine retention, sedation Age, weight, height and body mass index, duration of pregnancy, parity and gravity

ELIGIBILITY:
Inclusion Criteria:

* full-term, singleton, pregnant women,
* aged 18-35 years,
* scheduled for elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical class III or more
* multiple gestation.
* Patients with a history of allergy to any of the study drugs, ,
* coagulopathy,
* local infection,
* history of chronic pain or
* regular opioid use;
* inability to comprehend the numeric pain scale (NRS);
* and requirement for conversion to general anesthesia after spinal anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 15 minutes after intervention till 24 hours after suregery
  hours

SECONDARY OUTCOMES:
numeric pain scale | at 0.5, 1, 2, 4, 6, 18, 24 hours postoperative
  from 0-10
postoperative morphine requirement | 15 minutes after intervention till 24 hours after surgery
  mg
time to independent movement | 15 minutes after intervention till 24 hours after surgery
  hours
obstetric quality-of-recovery score | 24 hours after surgery
  grade the following 0-10: Moderate pain Severe pain Nausea or vomiting Feeling dizzy Shivering Have been comfortable Able to mobilise independently Can hold baby without assistance Can feed/nurse baby without assistance Can look after personal hygiene/toilet Feeling in control
opioid related complication | 24 hours after surgery
  nausea, vomiting, itching, urine retention, sedation

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available from the PI upon reasonable request